CLINICAL TRIAL: NCT06632444
Title: A Randomised, Double-blind, Placebo-controlled, Multicentre, Phase III Trial Evaluating Long-term Efficacy and Safety of Survodutide Weekly Injections in Adult Participants With Noncirrhotic Non-alcoholic Steatohepatitis/Metabolic Dysfunction-associated Steatohepatitis (NASH/MASH) and (F2) - (F3) Stage of Liver Fibrosis
Brief Title: LIVERAGE™: A Study to Test Whether Survodutide Helps People With a Liver Disease Called NASH/MASH Who Have Moderate or Advanced Liver Fibrosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1404-0044; 2024-513739-25-00 (Registry Identifier: CTIS); U1111-1306-9071 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Dysfunction Associated Steatohepatitis (MASH); Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Survodutide (Experimental)
  Interventions: Drug: Survodutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Survodutide — Subcutaneous injection
  Other Names: BI 456906
  Arms: Survodutide
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
This study is open to adults who are at least 18 years old living with obesity and have:

* a confirmed liver disease called non-alcoholic steatohepatitis (NASH)/metabolic associated steatohepatitis (MASH) and
* moderate or advanced liver fibrosis

People with a history of acute or chronic liver diseases other than MASH or chronic alcohol intake cannot take part in this study. The purpose of this study is to find out whether a medicine called survodutide helps people with MASH and moderate or advanced liver fibrosis improve their liver function.

This study has 2 parts. The purpose of the first part of this study is to find out the effect of survodutide on MASH and liver fibrosis. The purpose of the second part is to find out how safe and effective survodutide is in improving liver function. Participants are put into 2 groups randomly, which means by chance. 1 group gets survodutide and 1 group gets placebo. Placebo looks like survodutide but does not contain any medicine. Each participant has twice the chance of getting survodutide. Participants and doctors do not know who is in which group. Participants inject survodutide or placebo under their skin once a week. The survodutide doses are slowly increased until the target dose is reached. All participants receive counselling to make changes to their diet and to exercise regularly.

Participants are in the study for up to 7 years. During this time, they regularly visit the study site or have remote visits by video call. For about the first year of the study, participants have these visits every 2 weeks, increasing to every 4 weeks and then every 6 weeks. After being in the study for a little over a year participants will then alternate between visiting the study site or having a remote visit every 3 months until the end of the study.

The doctors check participants' health and take note of any unwanted effects. The participants' body weight and effects on the stomach and intestines are regularly measured. At some visits the liver is measured using different imaging methods. At 2 or 3 visits doctors take a small sample of liver tissue (biopsy). The participants also fill in questionnaires about their symptoms and quality of life. The results are compared between the groups to see whether the treatment works.

ELIGIBILITY:
Inclusion criteria:

1. Male or female participants ≥18 years (or who are of legal age in countries where that is greater than 18 years) of age at time of consent
2. Diagnosis of MASH (non-alcoholic fatty liver disease (NAFLD)) activity score [NAS] ≥4
3. Stable body weight defined as less than 5% self-reported change in body weight 3 months prior to the screening or during the period between the historical biopsy and randomisation, if a historical biopsy is used
4. Be willing to maintain a stable diet and physical activity levels throughout the entire trial Further inclusion criteria apply

Exclusion criteria:

1. Any of the following liver laboratory test abnormalities at screening:

   * Serum AST and/or alanine aminotransferase (ALT) elevation ≥5x upper limit of normal (ULN)
   * Platelet count <140 000/mm^3 (<140 GI/L)
   * Alkaline phosphatase >2x upper limit of normal (ULN)
   * Abnormal synthetic liver function as defined by screening central laboratory evaluation:

     * Albumin below <3.5 g/dL (35.0 g/L)
     * OR International normalised ratio (INR) of prothrombin time >1.3
     * OR total serum bilirubin concentration ≥1.5x ULN
2. Any history or evidence of acute or chronic liver disease other than MASH
3. Histologically documented liver cirrhosis (fibrosis stage F4), either at screening or in a historical biopsy
4. History of or current diagnosis of hepatocellular carcinoma
5. History of or planned liver transplant
6. Inability or unwillingness to undergo a liver biopsy at screening (if a suitable historical biopsy is unavailable for central review), or during trial conduct.
7. History of portal hypertension or presence of decompensated liver disease
8. Model for end-stage liver disease (MELD) score ≥12 due to liver disease. Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2031-12-27 (Estimated); Study Completion 2031-12-27 (Estimated)

PRIMARY OUTCOMES:
Part 1: Resolution of MASH without worsening of liver fibrosis on MASH Clinical Research Network (CRN) fibrosis score | Baseline and at Week 52.
Part 1: At least a 1-point improvement in fibrosis stage with no worsening of MASH | Baseline and at Week 52.
Part 2: Time to first occurrence of any of components of the composite endpoint consisting of progression to cirrhosis, all-cause mortality, liver transplant, hepatic decompensation event(s), worsening of MELD score to ≥15, progression to CSPH | Up to 7 years.
  Progression to cirrhosis is defined as histological fibrosis score CRN F4. MELD = Model for End-stage Liver Disease CSPH =clinically significant portal hypertension

SECONDARY OUTCOMES:
Key secondary endpoint part 1: Percentage change from baseline in body weight [kg] | Baseline and at Week 52.
Key secondary endpoint part 1: Absolute change from baseline in glycosylated haemoglobin (HbA1c) [%] | Baseline and at Week 52.
  This endpoint is specified only for the participants with type 2 diabetes mellitus.
Key secondary endpoint part 1: Absolute change from baseline in enhanced liver fibrosis (ELF) score | Baseline and at Week 52.
Key secondary endpoint part 1: Absolute change from baseline in liver stiffness [kPa] assessed by vibration-controlled transient elastography (VCTE) | Baseline and at Week 52.
Key secondary endpoint part 1: Achievement of no progression of fibrosis assessed by central pathology (yes/no) | Baseline and at Week 52.
Key secondary endpoint part 2: Percentage change from baseline in body weight [kg] | At baseline and at Week 114
Key secondary endpoint part 2: Absolute change from baseline in HbA1c [%] | At baseline and at Week 114
  This endpoint is specified only for the participants with type 2 diabetes mellitus.
Key secondary endpoint part 2: Absolute change from baseline in ELF score | At baseline and at Week 114.
Key secondary endpoint part 2: Absolute change from baseline in liver stiffness [kPa] assessed by VCTE | At baseline and at Week 114.
Key secondary endpoint part 2: Achievement of no progression of fibrosis assessed by central pathology (yes/no) | At baseline and at 7 years.
Key secondary endpoint part 2: Occurrence of all-cause hospitalisation (first and recurrent) | Up to 7 years.
Key secondary endpoint part 2: Time to first occurrence of any of the adjudicated components of the composite endpoint 5-point major adverse cardiac event (5P-MACE)5-point major adverse cardiac event (5P-MACE) | Up to 7 years.
Part 1: Improvement of liver fat content (LFC) | At baseline and at Week 52.
  Defined as at least 30% relative reduction in LFC compared with baseline assessed by Magnetic resonance imaging proton density fat fraction (MRI-PDFF).
  This endpoint will be reported only for a subset of participants in the MRI sub-study.
Part 2: Improvement of LFC | At baseline and at Week 114.
  Defined as at least 30% relative reduction in LFC compared with baseline assessed by MRI-PDFF.
  This endpoint will be reported only for a subset of participants in the MRI sub-study.
Part 1: Absolute change from baseline in LFC [%] in MRI-PDFF | At baseline and at Week 52.
  This endpoint will be reported only for a subset of participants in the MRI sub-study.
Part 2: Absolute change from baseline in LFC [%] in MRI-PDFF | At baseline and at Week 114.
  This endpoint will be reported only for a subset of participants in the MRI sub-study.
Part 1: Absolute change from baseline in alanine aminotransferase (ALT) [U/L] | At baseline and at Week 52.
Part 2: Absolute change from baseline in alanine aminotransferase (ALT) [U/L] | At baseline and at Week 114.
Part 1: Absolute change from baseline in aspartate aminotransferase (AST) [U/L] | At baseline and at Week 52.
Part 2: Absolute change from baseline in aspartate aminotransferase (AST) [U/L] | At baseline and at Week 114.
Part 1: Absolute change from baseline in systolic blood pressure (SBP) [mmHg] | At baseline and at Week 52.
Part 2: Absolute change from baseline in systolic blood pressure (SBP) [mmHg] | At baseline and at Week 114.
Part 1: Absolute change from baseline in diastolic blood pressure (DBP) [mmHg] | At baseline and at Week 52.
Part 2: Absolute change from baseline in diastolic blood pressure (DBP) [mmHg] | At baseline and at Week 114.
Part 1: Absolute changes from baseline in lipids [mg/dL] (including but not limited to: total cholesterol, LDL cholesterol, very low-density lipoprotein [VLDL] cholesterol, high-density lipoprotein [HDL] cholesterol, triglycerides) | At baseline and at Week 52.
  LDL=low-density lipoprotein
Part 2: Absolute changes from baseline in lipids [mg/dL] (including but not limited to: total cholesterol, LDL cholesterol, very low-density lipoprotein [VLDL] cholesterol, high-density lipoprotein [HDL] cholesterol, triglycerides) | At baseline and at Week 114.
Part 1: Absolute change from baseline in free fatty acids [mg/dL] | At baseline and at Week 52.
Part 2: Absolute change from baseline in free fatty acids [mg/dL] | At baseline and at Week 114.
Part 1: Progression to cirrhosis (defined as histological fibrosis score CRN F4) (yes/no) | At baseline and at Week 52.

CONTACTS AND LOCATIONS:
Locations (507):
- United States (159):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Institute for Liver Health II DBA Arizona Clinical Trials, Peoria, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Arizona Liver Health - Tucson, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Velocity Clinical Research-Chula Vista, Chula Vista, California
  - Southern California Research Center, Coronado, California
  - Velocity Clinical Research-Gardena-69773, Gardena, California
  - Velocity Clinical Research-Huntington Park, Huntington Park, California
  - 310 Clinical Research, Inglewood, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Om Research, LLC, Lancaster, California
  - ARK Clinical Research, Long Beach, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Catalina Research Institute, LLC - Montclair, Montclair, California
  - Velocity Clinical Research - Boise, North Hollywood, California
  - Clinnova Research Solutions, Orange, California
  - Fomat Medical Research, Oxnard, California
  - California Liver Research Institute, Pasadena, California
  - Cadena Care Institute, Llc, Poway, California
  - Ficramed Research Institute, Poway, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Metro Clinical Trials, San Bernardino, California
  - Acclaim Clinical Research, San Diego, California
  - Velocity Clinical Research, Santa Ana, Santa Ana, California
  - Om Research, LLC, Victorville, California
  - Future Innovative Treatments, Colorado Springs, Colorado
  - South Denver Gastroenterology PC, Englewood, Colorado
  - Connecticut Gastroenterology Clinical Research Foundation, Bristol, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Synergy Healthcare, Brandon, Florida
  - Access research Institute, Brooksville, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - K2 Medical Research, Clermont, Florida
  - Hi Tech and Global Research, LLC, Coral Gables, Florida
  - Top Medical Research, Inc, Cutler Bay, Florida
  - Covenant Metabolic Specialists, LLC - Fort Myers, Fort Myers, Florida
  - Neoclinical Research, Hialeah, Florida
  - Evolution Clinical Trials, Hialeah Gardens, Florida
  - Global Research Associates, Homestead, Florida
  - Lake Center for Clinical Research, Lady Lake, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - K2 Medical Research, Maitland, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - Optimus U Corporation-Miami-69452, Miami, Florida
  - Schiff Center Liver Diseases, Miami, Florida
  - BioMed Research & Medical Center, Miami, Florida
  - ECIR Miami Holdings LLC dba IMIC, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - GI Pros Research, Naples, Florida
  - Charter Research, Orlando, Florida
  - K2 Medical Research, Orlando, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - Endoscopic Research, Inc, Orlando, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - MplusM - Best Choice Medical and Research Service, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Metabolic Specialist, LLC - Riverview, Riverview, Florida
  - Global Clinical Professionals, St. Petersburg, Florida
  - Synergy Healthcare, St. Petersburg, Florida
  - International Center for Research, Tampa, Florida
  - Charter Research, The Villages, Florida
  - Covenant Metabolic Specialists, LLC - University Park, University Park, Florida
  - Conquest Research, Winter Park, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - EmVenio Research Center at Prime Healthcare- Atlanta, Riverdale, Georgia
  - ASHA Clinical Research - Munster, LLC, Hammond, Indiana
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas Medical Clinic PA, Topeka, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Clinton Township, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - MNGI Digestive Health, PA, Minneapolis, Minnesota
  - Gastrointestinal Associates, PA, Flowood, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - ObjectiveHealth-GI Associates Research, Columbia, Missouri
  - Kansas City Gastroenterology & Hepatology Physicians Group, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Jubilee Clinical Research, Inc, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - IMA Clinical Research-Warren-69742, Warren Township, New Jersey
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Basil Clinical, Laurelton, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - Carolina Researche, Greenville, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Columbus Clinical Research Inc., Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - ObjectiveHealth-DSI Research, Springboro, Ohio
  - Northshore Gastroenterology Research, Westlake, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - US Digestive Health, Flourtown, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - US Digestive Health, Lancaster, Pennsylvania
  - US Digestive Health, Wyomissing, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - ObjectiveHealth-Columbia Digestive Health Research, Columbia, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Premier Medical Group, Clarksville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - IMA Clinical Research Austin, Austin, Texas
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - Velocity Clinical Research, Austin, Austin, Texas
  - Bellaire Clinical Research, LLC, Bellaire, Texas
  - South Texas Research Institute-Brownsville-68426, Brownsville, Texas
  - Epic Medical Research - Carrollton, Carrollton, Texas
  - Pinnacle Clinical Research - Corpus Christi, Corpus Christi, Texas
  - Velocity Clinical Research-Dallas-69170, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Soma Clinical Trials, Denison, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - South Texas Research Institute-Edinburg-67012, Edinburg, Texas
  - EmVenio Research Center at Prime Healthcare, Farmers Branch, Texas
  - Care United Research, Forney, Texas
  - Epic Medical Research - Garland, Garland, Texas
  - Pinnacle Clinical Research, LLC, Georgetown, Texas
  - HRI Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Research Physicians Network, Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - GI Alliance, Mansfield, Texas
  - Biopharma Informatic LLC, McAllen, Texas
  - Centex Studies, Inc., McAllen, Texas
  - North Texas Research Institute - Dallas, Mesquite, Texas
  - Epic Medical Research - Plano, Plano, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - American Research Corporation, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Pinnacle Clinical Research, LLC, San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - HASresearch, San Antonio, Texas
  - Velocity Clinical Research, Waco, Waco, Texas
  - Objective Health-Digestive Research of Central Texas, Waco, Texas
  - ObjectiveHealth-Digestive Health Research of North Texas, Wichita Falls, Texas
  - Liver Institute of Virginia-Bremo, Newport News, Virginia
  - GI Select Health Research LLC, Richmond, Virginia
  - Medical College of Virginia Hospitals, Richmond, Virginia
  - Velocity Clinical Research-Seattle-69881, Seattle, Washington
  - Velocity Clinical Research-Spokane-69716, Spokane, Washington
- Argentina (11):
  - CIPREC, Buenos Aires
  - IDIM - Instituto de Diagnostico e Investigaciones Metabolicas, Buenos Aires
  - Buenos Aires Macula S.A., Buenos Aires
  - Mautalen- Salud e Investigacion, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Glenny Corp - Centro Médico Saavedra, Buenos Aires
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma Buenos Aires
  - Hospital Universitario Austral, Pilar
  - DIM Clinica Privada, Ramos Mejía
  - Hospital El Cruce, San Juan Bautista
- Australia (9):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (6):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Ordensklinikum Linz GmbH, Linz
  - Klinik Landstrasse, Vienna
  - AKH - Medical University of Vienna, Vienna
  - Hospital Hietzing, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (7):
  - ULB Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
  - Roeselare - HOSP AZ Delta, Roeselare
- Brazil (10):
  - Universidade Federal do Rio de Janeiro, Barra
  - Hospital Universitário João de Barros Barreto, Belém
  - Hospital das Clinicas da Universidade Federal de Minas Gerais (HCUFMG), Belo Horizonte
  - Universidade Estadual Paulista 'Julio De Mesquita Filho', Botucatu
  - Centro de Pesquisa Clinica do Brasil Ltda, Brasília
  - Hospital das Clinicas da Faculdade de Medicina da USP, Cerqueira César
  - Hospitalar Moinhos de Vento, Porto Alegre
  - Universidade Federal do Rio Grande do Sul, Porto Alegre
  - Hospital de Base - Fac Med de Sao Jose do Rio Preto, São José do Rio Preto
  - Rocco E Nazato Servicos Medicos LTDA, Vila Nova Conceição
- Bulgaria (7):
  - MHAT Sv. Ivan Rilski EOOD, Gorna Oryahovitsa
  - Multi-profile Hospital For Active Treatment-Uni Hospital Ltd., Panagyurishte
  - Acibadem City Clinic Tokuda University Hospital EAD, Sofia
  - Diagnostic Consultative Center Alexandrovska, Sofia
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski EAD, Sofia
  - Medical Military Academy MHAT Sofia, Sofia
  - Medical Center New Rehabilitation Center EOOD, Stara Zagora
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Pacific Gastroenterology Associates, Vancouver, British Columbia
  - Viable Clinical Research, Bridgewater, Nova Scotia
  - Toronto Liver Centre, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Centre de Médecine Métabolique de Lanaudière, Terrebonne, Quebec
  - Diex Recherche Québec, Québec
- Chile (3):
  - Edificio Fleming, La Serena
  - Centro de Investigaciones Médicas UC, Santiago
  - Centro de Investigaciones Clinicas Viña del Mar, Viña del Mar
- China (53):
  - Beijing Ditan Hospital Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Provincial People's Hospital, Changsha
  - Changzhou Third People's Hospital, Changzhou Shi
  - Chongqing Three Gorges Central Hospital, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangzhou Eighth People's Hospital,Guangzhou Medical University, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou
  - NanFang Hosptial, Guangzhou
  - The third affiliated hospital of Sun Yat-Sen University, Guangzhou
  - Guizhou People's Hospital, Guiyang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - The First hospital of Jiaxing, Jiaxing
  - Liaocheng People's Hospital, Liaocheng
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - The Second Hospital of Nanjing, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Ningbo Second Hospital, Ningbo
  - General Hospital of Ningxia Medical University, Ningxia
  - Pingxiang People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Renji Hospital Shanghai Jiaotong Univesrity School of Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - The Sixth People's Hospital of Shenyang, Shenyang
  - The Fifth People's Hospital of Suzhou, Suzhou
  - Tianjin Third Central Hospital, Tianjin
  - Tianjin Second People's Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi No. 5 People's Hospital, Wuxi
  - Second Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
  - Yanbian University Hospital, Yanji
  - Yueyang Central Hospital, Yueyang
  - Yuncheng Center Hopsital - West Compus, Yuncheng
  - Sixth People's Hospital of Zhengzhou, Zhengzhou
  - The Third People's Hospital of Zhenjiang, Zhenjiang
- Czechia (3):
  - Krajska nemocnice Liberec a.s., Liberec
  - Research Site s.r.o., Pilsen
  - General Faculty Hospital, Prague, Prague
- France (14):
  - CHU Amiens-Picardie, Amiens
  - Centre Hospitalier Universitaire D'Angers, Angers
  - Hôpital Beaujon, Clichy
  - HOP Dijon-Bourgogne, Côte-d'Or
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier De Versailles, Le Chesnay
  - Hopital De La Croix-Rousse, Lyon
  - Hôpital de l'Archet, Nice
  - Hôpital Claude Huriez, Nord-Pas-de-Calais
  - Hopitaux Universitaires Pitié-Salpétrière, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Universitaire De Bordeaux, Passec
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Rangueil - CHU de Toulouse, Toulouse
- Georgia (2):
  - Ltd "Health", Batumi
  - ISR-GEO Med Res Clin Healthycore, Tbilisi
- Germany (17):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH, Bochum
  - Universitätsklinikum Köln (AöR), Cologne
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universität des Saarlandes, Homburg
  - Eugastro GmbH, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
  - St. Josefs-Hospital Wiesbaden, Wiesbaden
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Hungary (4):
  - Dr. Rethy Pal Hospital, Békéscsaba
  - Obudai Egeszegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem Sebeszeti, Transzplantacios es Gasztroenterologiai Klinika, Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
- India (16):
  - Aryav Superspeciality Hospital, Ahemdabad
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Osmania Medical College & Hospital, Hyderabad, Afzalgunj
  - SR Kalla Memorial Hospital, Jaipur
  - ManglamPlus Medicity Hospital, Jaipur
  - G S V M, Kanpur, Kanpur
  - Atharva Multispecialty Hospital and research Centre, Lucknow
  - Practice Dr Kiranpal Singh, Mohali
  - Midas Multispeciality Hospital Pvt Ltd, Nagpur
  - Insitute of Liver and Billiary Sciences, New Delhi
  - All India Institute of Medical Sciences, New Delhi
  - Pandit Bhagwat Dayal Sharma Post Graduate Institute of Medical Sciences, Rohtak
  - Yashoda Hospitals - Secunderabad, Secunderabad
  - Surat Institute of Digestive Sciences, Surat
  - BAPS Pramukh Swami Hospital, Surat
  - Gujarat Gastro and Vascular Hospital, Surat
- Italy (11):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Az.Osp. Universitaria "Ospedali Riuniti", Foggia
  - Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Università degli Studi di Genova, Modena
  - Ospedale Maggiore della Carità, Novara
  - Policlinico "Paolo Giaccone", Palermo
  - Fondazione Policlinico Universitario Campus Bio-medico, Roma
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Ospedale "Casa Sollievo della Sofferenza", San Giovanni Rotondo
  - Universita Degli Studi di Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (54):
  - Fujita Health University Hospital, Aichi, Toyoake
  - The University of Tokyo Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Japan Institute for Health Security National Kohnodai Medical Center, Chiba, Ichikawa
  - Ehime University Hospital, Ehime, Toon
  - Fukuiken Saiseikai Hospital, Fukui, Fukui
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kurume University Hospital, Fukuoka, Kurume
  - Gifu Municipal Hospital, Gifu, Gifu
  - Nagano Municipal Hospital, Hanishina-gun
  - Hiroshima Red Cross Hospital and Atomic-bomb Survivors Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Sapporo Kosei General Hospital, Hokkaido, Sapporo
  - Japan Community Health Care Organization Hokkaido Hospital, Hokkaido, Sapporo
  - Hyogo College of Medicine Hospital, Hyogo, Nishinomiya
  - Tokyo Medical University Ibaraki Medical Center, Ibaraki, Inashiki-gun
  - Tokai University Hospital, Isehara
  - Kanazawa University Hospital, Ishikawa, Kanazawa
  - Shimane University Hospital, Izumo
  - Kagoshima University Hospital, Kagoshima, Kagoshima
  - Shin-yurigaoka General Hospital, Kanagawa, Kawasaki
  - St. Marianna University Hospital, Kawasaki-shi
  - Kagawa University Hospital, Kita-gun
  - Kobe University Hospital, Kobe
  - Kumamoto University Hospital, Kumamoto
  - Kumamoto Shinto General Hospital, Kumamoto, Kumamoto
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Japanese Red Cross Musashino Hospital, Musashino
  - Shinshu University Hospital, Nagano, Matsumoto
  - Nagasaki Medical Center, Nagasaki, Omura
  - Nara Medical University Hospital, Nara, Kashihara
  - Niigata University Medical and Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka City University Hospital, Osaka, Osaka
  - Oita Cardiovascular Hospital, Ōita
  - Saga University Hospital, Saga
  - Osaka Rosai Hospital, Sakai
  - Seichokai Bell Land General Hospital, Sakai
  - Sendai Tokushukai Hospital, Sendai
  - JCHO Shimonoseki Medical Center, Shimonoseki
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Juntendo University Shizuoka Hospital, Shizuoka, Izunokuni
  - Suita Hospital, Suita-Shi
  - The University of Osaka Hospital, Suita-shi
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi
  - Institute of Science Tokyo Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Toranomon Hospital, Tokyo, Minato-ku
  - Mie University Hospital, Tsu
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama City University Hospital, Yokohama
- Jordan (2):
  - The Speciality Hospital (TSH), Amman
  - Jordan University Hospital, Jordan
- Kazakhstan (2):
  - Institute of Gastroenterology, Gepatology and Metabolism LLP, Almaty
  - Asfendiyarov Kazakh National Medical University, Almaty
- Malaysia (4):
  - Hospital Ampang, Ampang
  - Hospital Universiti Sains Malaysia, Kota Bharu
  - University of Malaya Medical Centre, Kuala Lumpur
  - Queen Elizabeth Hospital, Putrajaya
- Mexico (8):
  - Centro de Investigacion Clinica del Pacifico (CICPA), Acapulco de Juárez
  - Clinicos Asociados BOCM SC, Benito Juarez, Mexico
  - Centro de Investigación y Gastroenterología, Col. Xoco
  - Instituto de Diabetes, Obesidad y Nutrición S.C., Cuernavaca
  - Centro de Investigación y Gastroenterología, Mexico City
  - Medical Care and Research, Mérida
  - Practice Dr Rosa Isela Luna Ceballos, Veracruz
  - Centro de Alta Especialidad del Estado de Veracruz, Xalapa
- Netherlands (3):
  - Amsterdam UMC Locatie VUMC, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam
  - Franciscus Gasthuis, Rotterdam
- New Zealand (4):
  - New Zealand Clinical Research (NZCR), Grafton, Auckland
  - Middlemore Hospital, Papatoetoe, Auckland
  - Christchurch Hospital, Christchurch, Canterbury
  - Waikato Hospital, Hamilton, Waikato Region
- Poland (9):
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Santa SP. z o.o, Lodz
  - FutureMeds Lodz, Lodz
  - Uniwersytecki Szpital Kliniczny Nr 1 W Lublinie, Lublin
  - ID Clinic, Mysłowice
  - FutureMeds Warszawa Centrum, Warsaw
  - Bodyclinic sp. z o.o. sp.k., Warsaw
  - FutureMeds Wroclaw, Wroclaw
  - EMC Instytut Medyczny S.A. - Wroclaw, Wroclaw
- Puerto Rico (3):
  - Klinical Investigations Group, LLC, San Juan
  - Latin Clinical Trial Center, San Juan
  - FDI Clinical Research, San Juan
- Romania (6):
  - Arensia Clinics S.R.L., Bucharest
  - Cluj Napoca Clinical County Hospital, Cluj-Napoca
  - Regional Institute of Gastroenterology Hepatology "Prof. Dr. O. Fodor", Cluj-Napoca
  - Spitalul Clinic Judetean De Urgenta Craiova, Craiova
  - Gastromedica Srl, Iași
  - Spital Judetean De Urgenta Satu Mare, Satu Mare
- Saudi Arabia (2):
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - King Abdulaziz Medical City, National Guard Health Affairs, Riyadh
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore
- South Africa (3):
  - Lenasia Clinical Trial Centre, Johannesburg
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
  - Inspired GI Care, Plumstead
- South Korea (12):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Deagu
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico de Santiago, Santiago de Compostela
- Switzerland (4):
  - Fondazione Epatocentro Ticino, Arzo
  - University Hospital Bern, Bern
  - Hopitaux Universitaires de Geneve (HUG), Geneva
  - University Hospital Zurich, Zurich
- Taiwan (11):
  - Chang-Hua Christian Hospital, Changhua
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsuing City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation (CGMF) - Linkou Bran, Taoyuan
- Turkey (Türkiye) (8):
  - Ankara Üniversitesi Tıp Fakültesi Hastanesi, Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Uludag Universitesi Tip Fakultesi, Bursa
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Fatih
  - Koc Universitesi Hastanesi, Istanbul
  - Memorial Bahçelievler Hospital, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Recep Tayyip Erdogan Universitesi Egitim ve Arastirma Hastanesi, Rize
- United Kingdom (21):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Velocity Clinical Research, Bristol, Bristol
  - Elpida Clinical Trials - Edgware Community Hospital, Edgware
  - Panthera Biopartners - North London, Enfield
  - Frimley Park Hospital NHS Foundation Trust, Frimley
  - Panthera Biopartners - Glasgow, Glasgow
  - Royal Free Hospital, London
  - King's College Hospital, London
  - Chelsea and Westminster Hospital NHS Foundation Trust - Chelsea and Westminster Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Accellacare North London, Northwood
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Accellacare - Orpington, Orpington
  - Panthera Biopartners - Preston, Preston
  - Panthera Biopartners - Manchester, Rochdale
  - Panthera Biopartners - Sheffield, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Elpida Sciences Clinical Trials, Wigan
  - Panthera Biopartners - York, York

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement '. For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com